CLINICAL TRIAL: NCT07286708
Title: Effect of a Serious Video Game Versus Traditional Training on Basic Life Support Knowledge and Skills in Adolescents: A Randomized Controlled Trial
Brief Title: Serious Game vs Traditional BLS Training in Adolescents
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Burcu SELVI CALSIKAN (Other)
Responsible Party: Sponsor-Investigator, Burcu SELVI CALSIKAN, Assistant Professor, Istanbul Arel University
Organization: Istanbul Arel University (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 2020/177
Record Dates: First submitted 2025-12-03; First posted 2025-12-16 (Actual); Last update posted 2025-12-17 (Actual); Status verified 2025-12

CONDITIONS: Basic Life Support Training Course; Cardiopulmonary Resuscitation (CPR)
Keywords: Adolescent; Basic life support; Traditional Training; Serious Video Game

STUDY DESIGN:
Intervention Model Description: Participants were randomly assigned to either the video game-based CPR training group or the traditional instructor-led CPR training group in a parallel two-arm design.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Video Game-Based CPR Training Group (Active Comparator): Participants in this arm received CPR training using the Lifesaver interactive video game developed by Resuscitation Council (UK). Training was completed individually under supervision using mobile phones. The video game provides a realistic CPR scenario and immediate feedback. No additional classical teaching was provided prior to the intervention.
  Interventions: Other: Lifesaver Video Game CPR Training
- Traditional Instructor-Led CPR Training Group (Active Comparator): Participants in this arm received traditional CPR training delivered by a certified instructor. Training included a theoretical lecture based on the Ministry of Health Adult Basic Life Support curriculum, followed by hands-on CPR practice using an adult manikin. Each session lasted approximately 2 hours. No video game or digital tool was used in this training.
  Interventions: Other: Traditional Instructor-Led CPR Training

INTERVENTIONS:
Other: Lifesaver Video Game CPR Training — The Lifesaver video game is an interactive, scenario-based CPR training tool developed by the Resuscitation Council (UK). Participants use their mobile phones to complete a simulated cardiac arrest scenario involving a teenage victim. The game teaches recognition of cardiac arrest, calling emergency services, performing chest compressions, rescue breaths, and AED use. Training was completed individually under supervision.
  Arms: Video Game-Based CPR Training Group
Other: Traditional Instructor-Led CPR Training — Participants received a traditional instructor-led CPR training consisting of a theoretical lecture based on the Ministry of Health Adult Basic Life Support guidelines and hands-on CPR practice using an adult manikin. Training lasted approximately 2 hours and did not include any digital or game-based components.
  Arms: Traditional Instructor-Led CPR Training Group

SUMMARY:
This randomized controlled trial aimed to compare the effects of a serious video game and traditional training on adolescents' basic life support (BLS) knowledge and skills. The study was conducted at Üsküdar High School in Istanbul, Turkey, between November 2021 and June 2022. Eleventh-grade students aged 15-17 years who had not previously received BLS training were randomly assigned to a video game group or a traditional education group. A total of 117 students completed the study (58 in the video game group and 55 in the traditional education group). The video game group received BLS education using the Lifesaver serious game, while the traditional group received a lecture based on national BLS guidelines and hands-on practice with a CPR training manikin. BLS knowledge and skills were assessed at baseline, 1 month, and 6 months using validated knowledge and skill assessment forms. The primary objective was to determine whether the serious game improved BLS knowledge and skill scores compared with traditional training and whether the effect persisted at 1- and 6-month follow-up.

DETAILED DESCRIPTION:
This randomized controlled trial evaluated the effectiveness of a serious video game compared with traditional training on adolescents' basic life support (BLS) knowledge and skills. A total of 117 high school students (aged 15-17 years) were randomly assigned to either the video game group (Lifesaver interactive scenario) or the traditional lecture-plus-practice group. All participants completed baseline, 1-month, and 6-month assessments using a 15-item BLS knowledge test and a 22-item skill performance checklist completed on a CPR manikin.

The video game group received a 13-minute interactive scenario-based BLS training, while the control group received a guideline-based lecture and hands-on manikin practice. Outcomes included changes in BLS knowledge and skill scores over time and group differences in short- and long-term retention.

Data were analyzed using nonparametric tests due to non-normal distribution. The study aimed to determine whether the serious game improves BLS learning and retention compared with traditional instruction.

ELIGIBILITY:
Inclusion Criteria:

* Students enrolled in the 11th grade at Üsküdar High School, Aged 15-17 years,
* Volunteered to participate in the study,
* Owns a smartphone capable of running the Lifesaver video game,
* No health problems affecting verbal communication,
* Provided written informed consent signed by both the student and their parent/guardian

Exclusion Criteria:

* Received Basic Life Support (BLS/CPR) training within the past 12 months,
* Transferred to another school during the study period,
* Declined to participate or withdrew consent at any time

Ages: 15 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 117 (Actual)
Dates: Start 2021-11-22 (Actual); Primary Completion 2022-06-17 (Actual); Study Completion 2022-12-02 (Actual)

PRIMARY OUTCOMES:
Change in CPR Knowledge Score After Training | Baseline, 1 month after training, and 6 months after training
  A multiple-choice CPR knowledge assessment consisting of 15 items was used to measure adolescents' theoretical understanding of adult Basic Life Support. Each correct answer was scored as 1 point, with total scores ranging from 0 to 15. Knowledge scores were measured at baseline (pre-test), 1 month after training, and 6 months after training in both groups. The primary outcome is the change in knowledge score from baseline to follow-up.

SECONDARY OUTCOMES:
Change in CPR Skill Performance Score After Training | Baseline, 1 month, and 6 months after training
  A 22-item CPR skill performance checklist scored using a 3-point Likert scale (0 = insufficient, 1 = needs improvement, 2 = sufficient), with total scores ranging from 0 to 44. Skill performance was assessed using an adult CPR manikin at baseline, 1 month, and 6 months after training. The outcome reflects changes in CPR skill competency over time.

CONTACTS AND LOCATIONS:
Locations (1):
- Istanbul Uskudar High School, Üsküdar, Istanbul, Turkey (Türkiye)

REFERENCES:
- See also: Related Info — https://life-saver.org.uk/